CLINICAL TRIAL: NCT06614621
Title: A Single-arm, Single-center, Prospective Clinical Study of Adebelimab Combined With Chemotherapy for First-line Treatment of Sequential Adebelimab Plus Apatinib Maintenance Therapy in Patients With Extensive-stage Small Cell Lung Cancer
Brief Title: A Study of Adebelimab Combined With Chemotherapy as a First-line Treatment Sequential Treatment for Extensive-stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJ-SCLC-01
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Extensive-Stage Small Cell Lung Cancer
Keywords: Adebrelimab; Apatinib Mesylate Tablets; Etoposide
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extensive-stage small cell lung cancer (Experimental): Therapeutic medications
  Interventions: Drug: Adebrelimab +Etoposide+Platinum-based drugs; Drug: Maintenance treatment period:

INTERVENTIONS:
Drug: Adebrelimab +Etoposide+Platinum-based drugs — Adebrelimab：20mg/kg或1200mg ivgtt ，d1 ，Q3W Etoposide injection (E): 100mg/m2, ivgtt, d1,d2,d3,Q3W Platinum-based drugs：75mg/m2， ivgtt， d1,d2,d3,Q3W
Drug: Maintenance treatment period: — Adebrelimab：20mg/kg或1200mg，IV, Q3W； Apatinib Mesylate Tablets：250mg，P.O，qod

SUMMARY:
A study of adebelimab in combination with chemotherapy in the first-line treatment of extensive-stage small cell lung cancer

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy (PFS, ORR, DCR, OS) and safety of adebelimab in combination with chemotherapy as a first-line treatment for the maintenance treatment of adebelimab plus Apatinib Mesylate Tablets with extensive-stage small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Patients with extensive-stage small cell lung cancer confirmed by pathological histology or cytology (excluding composite and small cell lung cancer);
2. Age at the time of signing the informed consent: 18-75 years old (including 18 years old and 75 years old), male or female;
3. United States Eastern Cooperative Oncology Group (ECOG) score performance status of 0 or 1;
4. Have not received prior systemic therapy for extensive-stage small cell lung cancer;
5. At least one measurable lesion per RECIST v1.1 criteria;
6. Expected survival ≥ 3 months;
7. Normal function of major organs, i.e., meeting the following criteria:

1) Routine blood test: hemoglobin (Hb) ≥90g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelets (PLT) ≥ 100×109/L; White blood cell count (WBC) ≥ 3.0×109/L; 2) Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (for patients with tumor liver metastasis, ≤5×ULN); Serum total bilirubin (TBIL) ≤ 1.5× ULN (Gilbert syndrome subjects, ≤3× ULN; In patients with liver metastases, total bilirubin ≤3× ULN); Serum creatinine (Cr) ≤ 1.5× ULN or creatinine clearance ≥ 50ml/min; 3) Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤1.5×ULN; 8. Females of childbearing potential should agree that contraception (such as intrauterine device [IUD], contraceptive pill or condom) must be used during the study and for 6 months after the end of the study; Negative serum pregnancy test within 28 days prior to study enrollment and must be non-lactating subjects; Males should be subjects who agree to use contraception for the duration of the study and for 6 months after the end of the study period.

9. Subjects voluntarily joined this study, signed the informed consent form, had good compliance, and cooperated with follow-up

Exclusion Criteria:

* 1. Known allergy to any of the drugs in the study; 2. Previous or concurrent other malignant tumors, excluding cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast (DCIS), papillary thyroid carcinoma and other malignant tumors that have been adequately treated and cured for ≥ 5 years before the first dose and have evidence to confirm that there is no recurrence and metastasis; 3. Presence of symptomatic or active central nervous system (CNS) metastases or carcinomatous meningitis (asymptomatic or post-treatment stable brain metastases are allowed); 4. Presence of active or previous autoimmune disease or immunodeficiency; 5. Presence of active or previous autoimmune disease or immunodeficiency Imaging (CT or MRI) shows tumor invasion of or ill-demarcation of large vessels; or judged by the investigator that the subject's tumor has a very high probability of invading important blood vessels and causing fatal hemorrhage during treatment; 6. Have hypertension that is not well controlled by antihypertensive medication (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 100 mmHg); 7. Cardiovascular and cerebrovascular diseases with significant clinical significance:

  * Cerebrovascular accident (excluding lacunar cerebral infarction, minor cerebral ischemia or transient ischemic attack, etc.), myocardial infarction, unstable angina, poorly controlled arrhythmia (including QTc interval ≥ 450 ms for males and ≥ 470 ms for females) within 6 months before the first dose of the study drug (QTc interval is calculated by Fridericia's formula);
  * United States New York Heart Association (NYHA) cardiac function class > class II or left ventricular ejection fraction (LVEF) <50%; 8. Active or uncontrolled severe infection;
  * Known human immunodeficiency virus (HIV) infection;
  * History of known clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must rule out active HBV infection, i.e., HBV DNA positive (>1×104 copies/mL or >2000 IU/ml);
  * Known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies/mL), or other hepatitis, cirrhosis; 9. Patients who are judged by the investigator to be accompanied by uncontrollable third space effusions such as pleural effusion, pericardial effusion or peritoneal effusion, which require puncture and drainage; or those who have received ascites and pleural effusion drainage within 14 days before the first dose; 10. Patients with interstitial pneumonia or interstitial lung disease, or a history of interstitial pneumonia or interstitial lung disease requiring hormonal therapy, or other pulmonary fibrosis, chronic pneumonia, pneumonia-induced by drugs or radiotherapy, history of congenital pneumonia, or any evidence of active pneumonia on chest CT scan that may interfere with the judgment of immune-related pulmonary toxicity; Patients with severe impairment of lung function confirmed by current pulmonary function tests; 11. Subjects who need to be treated with systemic corticosteroids (> 10 mg/day effective dose of prednisone) or other immunosuppressive medications within 14 days prior to the first dose or during the study. However, enrollment is allowed in the following cases: in the absence of active autoimmune disease, subjects are allowed to use topical or inhaled steroids and adrenal hormone replacement therapy at an effective dose of ≤ 10 mg/day prednisone; 12. Subject currently has any current disease or state that affects drug absorption, or subject cannot take apatinib orally; 13. Those whose urine routine shows that urine protein ≥2+, and the 24-hour urine protein quantification > 1.0g; 14. In the opinion of the investigator, the subject has any clinical or laboratory examination abnormalities or other reasons that make it unsuitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival（PFS） | 12 months
  First-line treatment with adebelimab plus chemotherapy for sequential adebelimab plus apatinib maintenance therapy for progression-free survival (PFS) in patients with extensive-stage small cell lung cancer

SECONDARY OUTCOMES:
Objective response rate（ORR） | 12 months
  Objective response rate (ORR) of adebelimab plus chemotherapy in first-line treatment of sequential adebelimab plus apatinib maintenance therapy in patients with extensive-stage small cell lung cancer
Disease control rate（DCR） | 12 months
  Disease control rate (DCR) of adebelimab plus chemotherapy in first-line treatment of sequential adebelimab plus apatinib maintenance therapy in patients with extensive-stage small cell lung cancer

IPD SHARING:
Plan to Share IPD: No